CLINICAL TRIAL: NCT06103630
Title: Efficacy of Oropharyngeal Exercises for Patients With Residual Obstructive Sleep Apnea Using Mandibular Advancement Device
Brief Title: Efficacy of Oropharyngeal Exercises for Patients With Obstructive Sleep Apnea Using Mandibular Advancement Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-ER-112-396
Record Dates: First submitted 2023-10-16; First posted 2023-10-27 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-10

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: Obstructive Sleep Apnea; Mandibular Advancement Device therapy; Oropharyngeal muscle training
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Mandibular advancement device
  Interventions: Other: Mandibular advancement device
- Intervention group (Experimental): Participants will received 1-2 times a week, 12-week-intervention of Oropharyngeal Exercises and Mandibular advancement device.
  Interventions: Other: Oropharyngeal Exercises; Other: Mandibular advancement device

INTERVENTIONS:
Other: Oropharyngeal Exercises — Oropharyngeal Exercises
  Arms: Intervention group
Other: Mandibular advancement device — Mandibular advancement device

SUMMARY:
Oropharyngeal muscle training has emerged as a novel adjunctive treatment approach, involving training of the swallowing muscle group and tongue muscles to prevent tongue collapse, reduce tongue base volume during sleep, and strengthen muscle tension.

Therefore, the objective is to assess changes in oropharyngeal muscle strength, ultrasonographic tongue morphology, severity of sleep related breathing interruptions, clinical symptoms, and correlations among these factors. Oropharyngeal muscle training for patients with residual OSA using MAD can significantly 1. increase muscle strength and endurance. 2. reduce the severity of sleep-related breathing interruptions. 3. decrease clinical symptoms. 4. improve tongue morphology.

DETAILED DESCRIPTION:
Background:

Obstructive Sleep Apnea (OSA) refers to recurrent upper airway blockages during sleep, leading to symptoms like snoring, 2 interrupted breathing causing micro-awakenings, daytime sleepiness, impaired concentration, and various chronic conditions. The Mandibular Advancement Device (MAD) is a treatment method for OSA, suitable for mild to moderate cases and CPAP noncompliance. However, clinical use of MAD sometimes falls short in comprehensively alleviating the clinical symptoms of obstructive sleep apnea. Therefore, oropharyngeal muscle training has emerged as a novel adjunctive treatment approach, involving training of the swallowing muscle group and tongue muscles to prevent tongue collapse, reduce tongue base volume during sleep, and strengthen muscle tension. This training aims to increase overall respiratory tract rigidity and improve muscle responsiveness during reduced blood oxygen levels.

Given that some patients do not achieve the expected outcomes after MAD therapy, whether oropharyngeal muscle training can enhance treatment effects becomes a research focus. Thus, this study aims to apply oropharyngeal muscle training to patients who have not achieved the anticipated results following MAD treatment. The objective is to assess changes in oropharyngeal muscle strength, ultrasonographic tongue morphology, severity of sleep related breathing interruptions, clinical symptoms, and correlations among these factors.

Methods:

Fifty diagnosed OSA patients using MAD and consenting to participate are recruited. Patients agreeing to undergo 12 weeks of oropharyngeal muscle training form the treatment group, while those not agreeing form the control group. The treatment group undergoes 12 weeks of training, with weekly in-person follow-ups for treatment intensity adjustment and home-based sessions (30 mins, 1-3 times/day, 3-5 days/week) for a total of 12 weeks. The control group continues MAD therapy. Both groups undergo evaluations of muscle strength and endurance, various sleep physiological tests, ultrasonographic imaging of the tongue and oropharynx, and sleep questionnaire tests before and after the 12- week training period.

Expected Outcomes:

1. Oropharyngeal muscle training may increase muscle strength and endurance.
2. Oropharyngeal muscle training may reduce the severity of sleep-related breathing interruptions.
3. Oropharyngeal muscle training may decrease clinical symptoms.
4. Oropharyngeal muscle training may improve tongue morphology.

ELIGIBILITY:
Inclusion Criteria:

* OSA patients
* Aged over 20 years
* Wearing MAD (The amount of MAD is at least 50% of the maximum amount that the patient can achieve.)

Exclusion Criteria:

* Body Mass Index (BMI) ≧ 35
* Pregnancy
* Severe obstructive or restrictive lung disease
* Exercise with high-risk cardiovascular disease
* History of central or peripheral neurological disease resulting in an inability to perform exercise prescriptions
* Musculoskeletal or psychological disorders that prevent the performance of exercise prescriptions
* Chronic illnesses that are ongoing or not yet controlled

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea -index | Baseline to 12 weeks
  Assessed using Polysomnography (PSG). The average apnea and hypopnea events per hour, oxygen saturation index and the snoring index will be obtained during the sleep test(PSG).

SECONDARY OUTCOMES:
Tongue muscle strength | Baseline to 12 weeks
  The maximal muscle strength of genioglossus muscles using The Iowa Oral Performance Instrument (IOPI) system, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA) (kPa)
Jaw strength | Baseline to 12 weeks
  Jaw strength will be measured using a 'handheld' dynamometer (MicroFET○R2, Hoggan Scientific, USA). The data will be presented in kilogram-weight. The minimum score is 0 and a higher score indicates stronger in jaw strength.
Tongue muscle endurance | Baseline to 12 weeks
  The endurance of the genioglossus muscles using The Iowa Oral Performance Instrument (IOPI) system, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA) (in seconds).
Tongue Muscle Thickness | Baseline to 12 weeks
  Sonography will be performed over the participant's neck region to assess the changes in tongue muscle thickness during normal breathing.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hsia Hung, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan